CLINICAL TRIAL: NCT07045428
Title: An Exploratory, Single-Arm, Open-label Study of Safety, Pharmacokinetics, Biodistribution and Dosimetry of 68Ga-GP-01 Injection in Participants With Solid Tumors
Brief Title: 68Ga-GP-01 Injection in Solid Tumors Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GrandPharma (China) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ST1530-1
Record Dates: First submitted 2025-06-12; First posted 2025-07-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor Malignancies
Keywords: radiopharmaceutical

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open label trial aimed at evaluating the safety, pharmacokinetics, biodistribution, dosimetry, and preliminary ability to detect metastatic disease of 68Ga-GP-01 injection in participants with solid tumors.
  This study contains two parallel cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental)
  Interventions: Drug: 68Ga-GP-01 Injection

INTERVENTIONS:
Drug: 68Ga-GP-01 Injection — A certain mass dose of 68Ga-GP-01 will be used in this study, and the radiation dose will be no more than, enabling all participants will receive a radiation dose of 5±2 mCi in the study.

SUMMARY:
A company named Chengdu Shetai Medical Technology Co., Ltd. is conducting a research study to test a new type of scan for detecting solid tumors in patients who are scheduled for surgery.

During the scan, the investigators will use a special experimental drug called 68Ga-GP-01 Injection, which is given through a vein (IV). This drug isn't yet approved by the TGA for this use.

The scan works by targeting a protein called FAP that's often found in high amounts in tumor tissues. FAP is mainly present in cells surrounding tumors, but sometimes in cancer cells themselves too - especially in certain cancers like ovarian, breast, pancreatic, and some sarcomas. Researchers think this could be useful for both diagnosis and potential future treatments.

The GP-01 molecule is combined with a radioactive material (Gallium-68) that shows up on PET scans - a special imaging technique that can spot cancer cells in the body.

Currently, CT scans are the most common way to check for tumors before surgery. A PET/CT machine combines both technologies - it can show both the structure of participant's organs (CT) and detect cancer cells that have absorbed the radioactive tracer (PET).

In this study, the investigators want to see if 68Ga-GP-01 works better than standard PET/CT scans at finding tumors. After participant's surgery, the investigators will compare our scan results with participant's pathology report (the most accurate way to diagnose cancer) to check how accurate our method was.

Important: This is NOT a treatment for participant's cancer - it's just testing a new way to detect tumors.

About 20 patients at 4 Australian hospitals will participate. If participant is willing to join, participant's involvement will last about 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Agreed to participate by providing a signed informed consent form and can comply with study-related procedures.
2. Male or female aged ≥ 18 years old.
3. Patients with solid tumors planned to undergo surgical resection or laparoscopic exploration and histopathology confirmation.
4. Available CT/MRI images of suspected metastatic regions of cohort 1 patients; available CT/MRI images of both primary and metastatic regions of cohort 2 patients. .
5. Be capable of receiving 18F-FDG PET/CT scan.
6. Adequate renal function as determined by a creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula).
7. Females of childbearing potential must have a negative pregnancy test.. Male and female participants of childbearing potential must use at least 2 highly effective forms of contraception, one of which must be a barrier method, or agree to remain abstinent for duration of study participation and for 3 months following Ga agent.

Exclusion Criteria:

1. Any PET scan done within 10 physical half-lives of the PET agent prior to planned administration of 68Ga-GP-01.
2. Exposure to any investigational agent within 4 weeks prior to the planned administration of 68Ga-GP-01.
3. Major surgery, any systemic anti-cancer therapy or radiotherapy within 4 weeks prior to planned administration of 68Ga-GP-01.
4. Past or current history of another malignancy, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least 3 years;
5. Co-morbidities (e.g., hydronephrosis, kidney failure, liver failure, systemic or local inflammatory or autoimmune diseases or other conditions) that in the opinion of the investigator could compromise patient safety and/or protocol objectives.
6. Planned antineoplastic therapies from time of consent to planned surgery or laparoscopic exploration.
7. Planning to participate in any drug or device clinical trial during the study period.
8. Has a known or suspected allergic reaction to any components of the formulation used in 68Ga-GP-01.
9. Contraindications to PET/CT scan.
10. Has a medical, psychological, or social condition that, in opinion of the investigators will make it difficult to comply study procedures.
11. Female participants who are pregnant or lactating.
12. Other reasons determined by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of 68Ga-GP-01 | Within Day3 after dose
  Number of participants with treatment emergent adverse event, with abnormal laboratory tests results and abnormal 12-lead electrocardiograms (ECGs) readings.

IPD SHARING:
Plan to Share IPD: No